CLINICAL TRIAL: NCT02296398
Title: Retrospective and Prospective Study of Long-term Use of Romidepsin in Patients
Brief Title: Long-term Use of Romidepsin in Patients With CTCL
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Joan Guitart, MD, Northwestern University
Other Study IDs: STU95649
Record Dates: First submitted 2014-10-02; First posted 2014-11-20 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — romidepsin; Maintenance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Romidepsin therapy: Patients who received romidepsin per standard of care practice or included in other clinical trials (when receiving romidepsin therapy).
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin — Received romidepsin per standard of care or through a clinical trial for more than one cycle
  Other Names: Maintenance therapy

SUMMARY:
Cutaneous T-cell lymphomas (CTCL) are a heterogeneous group of neoplasm of skin-homing T cells that includes Mycosis Fungoid (MF), which is the most common, Sézary syndrome (SS), the leukemia variant of MF, and other variants of CTCL which are less prevalent. Clinical manifestations and prognosis are highly variable. Improving the management of this incurable disease with limited toxicity is the main point of the current research. Romidepsin is a well-tolerated histone deacetylase inhibitor which has demonstrated activity against advanced stages of CTCL. In November 2009, it was approved by the US Food and Drug Administration (FDA) for the treatment of CTCL in patients who have received at least one prior systemic therapy. FDA-dose approved is 14 mg/m2 days 1, 8, 15 of a 21 day-cycle. It is said that it should be continued as long as the patient receives benefit and tolerates the drug. We experienced in our clinic that a long-term (>6 months) use of Romidepsin, even with spared doses allows patients to maintain disease in complete remission or under control without severe side effects. We aim to demonstrate how many patients have benefited of this maintenance therapy, and detect the side effects related to the long-term use of Romidepsin, as well as characterize those patients that can get benefit of this therapy.

DETAILED DESCRIPTION:
This project is a retrospective and prospective chart review of patients who present at Northwestern Medical Faculty Foundation clinic with the diagnosis of CTCL. It includes Mycosis Fungoid, Sézary Syndrome and other subtypes of CTCL, like Cytotoxic Cutaneous T-cell lymphomas. Those patients that received or will be prescribed per standard of care with romidepsin for at least 1 month (or at least more than 1 cycle of treatment) will be reviewed. We estimate that 50 patients could fit the criteria above, since the drug started to be prescribed in the Dermatology Clinic. Clinical information regarding diagnosis, stage, prior treatment received, and therapeutic response will be recorded. Blood parameters such as cell blood count, calcium, magnesium, potassium, and albumin at baseline and after treatment with romidepsin will be reviewed, and recorded if abnormalities are detected. Electrocardiogram changes will also be checked and recorded. All the information will be gathered in an excel spreadsheet in order to perform a descriptive analysis. We aim to assess the use of romidepsin as maintenance therapy and assess which schedule of treatment was most frequently used and associated with a better response with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Cutaneous T-cell Lymphoma who present to the Northwestern Medical Faculty Foundation Dermatology clinic between January 1, 2009 and December 31, 2014
* Stages with more than 20% of bosy surface area affected or higher for MF and SS, and other CTCL variants
* Patients treated with romidepsin
* Between 18 and 89 years

Exclusion Criteria:

* Patients under 18 and over 89 years
* Patients with the diagnosis of CTCL that did not received romidepsin as a treatment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records of patients with a diagnosis of cutaneous T-cell lymphoma that have presented to the Northwestern Medical Faculty Foundation Dermatology clinic, who receive romidepsin per standard of care practice will be reviewed. Retrospective chart reviews will be conducted for data collected between January 1, 2009 (when romidepsin was initially prescribed) to May 28, 2014. The prospective portion of the study will review chart data collected between May 29, 2014 and December 31, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Free disease time with maintenance therapy with romidepsin | 4 weeks
  By the time patient received the first cycle the clinical response will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Joan Guitart, MD, Principal Investigator — Northwestern Univeristy
Locations (1):
- Northwestern University Dermatology Department, Chicago, Illinois, United States